CLINICAL TRIAL: NCT06308952
Title: Atorvastatin Pretreatment in Cerebrovascular Events (APICES) After Flow Diverter Implantation: Protocol of a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Atorvastatin Pretreatment in Cerebrovascular Events (APICES) After Flow Diverter Implantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duan Chuanzhi (Other)
Responsible Party: Sponsor-Investigator, Duan Chuanzhi, Professor, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024SL0006
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cerebrovascular Event; Stent Stenosis; Ischemic Stroke; Hemorrhagic Stroke; Stent Thrombosis; Death, Brain; Endothelial Dysfunction
Keywords: Atorvastatin; Intracranial aneurysm; Flow-diverter devices; Stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Brain Death; Intracranial Aneurysm; Stroke | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement. Investigators, other blinded investigators, subjects, and sponsors will not have access to any information regarding group assignment or related documents pertaining to the trial drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): placebo (composed mainly of starch, Frontage Pharma, Jiangsu, China) 20mg orally once daily for 180 days
  Interventions: Drug: Atorvastatin 20mg
- Experimental group (Experimental): atorvastatin (Pfizer, New York, USA) 20mg orally once daily for 180 days
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — Eligible subjects screened will enter the pretreatment period (at least 24 hours) and be randomly assigned to the trial group (oral atorvastatin) or the control group (placebo) to start receiving the trial drug (20mg, qd). Additionally, the patient was started on basic dual anti-platelet (aspirin 75mg qd + clopidogrel 75mg qd/ticagrelor 45mg bid).
  Other Names: Lipitor

SUMMARY:
APICES trial is an investigator-initiated, multicenter, multicenter, randomized, double-blind, placebo-controlled clinical trial that plans to enroll 396 patients with a 1-year follow-up, including a neurovascular imaging examination [digital subtraction angiography (DSA), CT angiography (CTA) or magnetic resonance angiography (MRA)] at 6 months after index treatment. It was designed in compliance with the Declaration of Helsinki and the International Conference on Harmonization Good Clinical Practice guidelines. The study was approved by the Ethics Committee of Zhujiang Hospital of South Medical University (2024-KY-032-02) and registered at ClinicalTrials.gov (NCT06308952). The participants will be recruited from twelve advanced stroke centers in China.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a disastrous subtype of stroke, which is associated with high mortality and morbidity. With the advancement of endovascular techniques, flow diverter (FD) devices have emerged as a preventive treatment for unruptured intracranial aneurysms (UIAs). Although a series of studies have demonstrated that FDs can achieve high rates of aneurysmal occlusion, the safety of FDs remains a concern, with a non-negligible risk of complications (5%-12%). Furthermore, previously published studies have also confirmed that FDs have a significantly higher rate of in-stent stenosis (ISS) compared with conventional stents, which remains a clinical issue requiring attention and resolution. However, there are currently no guideline recommendations or clinical evidence available on how to prevent complications in patients with IA after undergoing FD implantation, apart from conventional dual antiplatelet therapy.

Elevated low-density lipoprotein cholesterol (LDLC) levels increase the risk of vascular events. Lipid-lowing treatment with β-Hydroxy β-methylglutaryl-CoA reductase inhibitors (such as statins) is a cornerstone in avoiding such events. Several studies indicate that the advantages of statins could surpass their traditional role in lowering cholesterol levels, encompassing a range of additional benefits known as pleiotropic effects. Those multiple effects include anti-inflammatory function, vasodilation, anticoagulation, platelet inhibition, and antioxidants. Although the clinical benefit of statin pretreatment has been clarified in carotid artery stenting, percutaneous coronary intervention, and abdominal aortic aneurysm repair, its effect on endovascular treatment of UIAs remains unclear.

Due to the pleiotropic benefits beyond lipid lowering, the effect of statin pretreatment may theoretically contribute to the reduction of cerebrovascular events after FD implantation. Nevertheless, there is currently a lack of high-quality clinical evidence supporting this hypothesis. Thus, we designed the atorvastatin pretreatment in cerebrovascular events (APICES) randomized controlled trial (RCT) to explore whether statin pretreatment is superior to placebo in patients undergoing FD treatment for UIAs.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 to 75 years old, male or non-pregnant female;
2. UIA diagnosed by CTA, MRA, or DSA;
3. Maximal aneurysmal diameter between 3 and 25mm;
4. Understands the nature of the procedure and provision of written informed consent;
5. Indications for FD implantation with or without adjunctive coiling;
6. Is willing to return to the investigational site for follow-up according to our protocol.

Exclusion criteria:

Patients will be excluded if they meet any of the following criteria:

1. Contraindications to atorvastatin treatment or known allergy to atorvastatin;
2. Pregnancy or lactation;
3. Presence of other vascular lesions (coronary artery disease, abdominal aortic aneurysm, intracranial atherosclerotic stenosis, arteriovenous malformation, dural arteriovenous fistula, Moyamoya disease, etc.);
4. Prolonged statin therapy (≥30 days) or prior indications for atorvastatin therapy according to the Chinese guidelines for lipid management (2023) 21;
5. Ruptured aneurysms or target aneurysm received previous operative or endovascular treatment;
6. Patient currently using drugs that interact with atorvastatin metabolism (including transporter inhibitors, cyclosporine, protease inhibitors, other lipid-lowering medications (such as fibrates, ezetimibe, pcsk9 inhibitor, etc.), antacids, erythromycin, cytochrome P450 enzyme, colchicine, etc.);
7. Patients diagnosed with multiple intracranial aneurysms who require treatment for two or more intracranial aneurysms within a one-year period;
8. The target aneurysm is non-saccular (dissecting, fusiform, pseudo, infectious, etc.)
9. Other situations that the researcher deems unsuitable for inclusion in the study (inability to receive anti-platelet or anticoagulant medication; allergy or contraindication for the use of FD alloy, history of life-threatening allergy to contrast dye, ect).
10. Patient was determined that intravenous general anesthesia or general anesthesia with tracheal intubation could not be tolerated.
11. Unwilling to be followed up or likely to have poor treatment compliance at initial screening;
12. Life expectancy less than 3 years;
13. Severe neurological deficit that renders the patient unable to live independently (modified Rankin score ≥4);
14. Enrollment in another trial.

Withdrawal criteria

In this trial, participants who have provided written informed consent but are unable to complete the entire study for any reason will be withdrawn. These circumstances include the following:

1. The participants voluntarily quit the trial for various reasons;
2. Occurrence of serious adverse events (SAEs). The study may be terminated by the participants, principal investigators, ethics committee, sponsor, or regulatory authorities based on ethical considerations;
3. Early termination of the process based on the investigator's judgment in order to prevent development of severe complications;
4. Significant deviation in implementation, or the subject failed to comply with the scheduled protocol;
5. Miss the follow-up due to changes in working/living places, or fortuitous accident (traffic accident, bone fracture, accidental death, ect.). Thus, close follow-up should be conducted to determine their relationship with the usage of FD and experimental drug;
6. Flawed or absence of informed consents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy endopoint | 1 year
  Patients without new-onset cerebrovascular events within 12 months:
  1. Any documented stroke (clinical and imaging): hemorrhage stroke (any intracranial hemorrhage subtype confirmed by CT scan) or ischemic stroke (neurological dysfunction more than 24 hours after onset or new acute cerebral infarction lesion confirmed by imaging);
  2. the incidence of significant in-stent stenosis (a narrowing of the FD diameter exceeding 50% without pre-existing significant artery stenosis detected by 12-month angiographic follow-up).

SECONDARY OUTCOMES:
Safety endpoint | 1 year
  1. muscle-related adverse events (excluding those due to exercise or trauma);
  2. digestive system adverse events (dyspepsia, unexplained abdominal pain, biliary colic, gastrointestinal bleeding);
  3. Newly diagnosed cancer, diabetes, neurocognitive disorders, cataracts;
  4. all-caused death;
  5. the incidence and the degree of ISS;
  6. incomplete aneurysm occlusion;
  7. new-onset in-stent thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, MD, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo B, Kang H, Zhang H, Li T, Liu J, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X. Pipeline Embolization device for intracranial aneurysms in a large Chinese cohort: factors related to aneurysm occlusion. Ther Adv Neurol Disord. 2020 Nov 2;13:1756286420967828. doi: 10.1177/1756286420967828. eCollection 2020. PMID 33224273
- [Result] Vergouwen MD, Jong-Tjien-Fa AV, Algra A, Rinkel GJ. Time trends in causes of death after aneurysmal subarachnoid hemorrhage: A hospital-based study. Neurology. 2016 Jan 5;86(1):59-63. doi: 10.1212/WNL.0000000000002239. Epub 2015 Nov 20. PMID 26590269
- [Result] Huang C, Ma G, Tong X, Feng X, Wen Z, Huang M, Xu A, Yuan H, Shi H, Lin J, Li C, Ge R, Huang J, Peng C, Zhu Y, Wang T, Huang C, Guo Z, Liang S, Su S, Zhang X, Li X, Liu A, Duan CZ. Comparison of Pipeline embolization device versus Tubridge embolization device in unruptured intracranial aneurysms: a multicenter, propensity score matched study. J Neurointerv Surg. 2024 May 6;17(5):467-474. doi: 10.1136/jnis-2024-021623. PMID 38719444
- [Result] Hanel RA, Cortez GM, Lopes DK, Nelson PK, Siddiqui AH, Jabbour P, Mendes Pereira V, Istvan IS, Zaidat OO, Bettegowda C, Colby GP, Mokin M, Schirmer CM, Hellinger FR, Given C, Krings T, Taussky P, Toth G, Fraser JF, Chen M, Priest R, Kan P, Fiorella D, Frei D, Aagaard-Kienitz B, Diaz O, Malek AM, Cawley CM, Puri AS, Kallmes DF. Prospective study on embolization of intracranial aneurysms with the pipeline device (PREMIER study): 3-year results with the application of a flow diverter specific occlusion classification. J Neurointerv Surg. 2023 Mar;15(3):248-254. doi: 10.1136/neurintsurg-2021-018501. Epub 2022 Mar 15. PMID 35292570
- [Result] Qi P, Tong X, Liang X, Xue X, Wu Z, Feng X, Zhang M, Jiang Z, Wang D, Liu A. Flow diversion for posterior circulation aneurysms: a multicenter retrospective study. Ther Adv Neurol Disord. 2023 Jun 8;16:17562864231176187. doi: 10.1177/17562864231176187. eCollection 2023. PMID 37324979
- [Result] Hanel RA, Cortez GM, Coon AL, Kan P, Taussky P, Wakhloo AK, Welch BG, Dogan A, Bain M, De Vries J, Ebersole K, Meyers PM; SCENT Investigator Group. Surpass Intracranial Aneurysm Embolization System Pivotal Trial to Treat Large or Giant Wide-Neck Aneurysms - SCENT: 3-year outcomes. J Neurointerv Surg. 2023 Nov;15(11):1084-1089. doi: 10.1136/jnis-2022-019512. Epub 2022 Nov 14. PMID 36375835
- [Result] Kang H, Zhou Y, Luo B, Lv N, Zhang H, Li T, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Liu J. Pipeline Embolization Device for Intracranial Aneurysms in a Large Chinese Cohort: Complication Risk Factor Analysis. Neurotherapeutics. 2021 Apr;18(2):1198-1206. doi: 10.1007/s13311-020-00990-8. Epub 2021 Jan 14. PMID 33447904
- [Result] Kallmes DF, Hanel R, Lopes D, Boccardi E, Bonafe A, Cekirge S, Fiorella D, Jabbour P, Levy E, McDougall C, Siddiqui A, Szikora I, Woo H, Albuquerque F, Bozorgchami H, Dashti SR, Delgado Almandoz JE, Kelly ME, Turner R 4th, Woodward BK, Brinjikji W, Lanzino G, Lylyk P. International retrospective study of the pipeline embolization device: a multicenter aneurysm treatment study. AJNR Am J Neuroradiol. 2015 Jan;36(1):108-15. doi: 10.3174/ajnr.A4111. Epub 2014 Oct 29. PMID 25355814
- [Result] Colby GP, Bender MT, Lin LM, Beaty N, Caplan JM, Jiang B, Westbroek EM, Varjavand B, Campos JK, Huang J, Tamargo RJ, Coon AL. Declining complication rates with flow diversion of anterior circulation aneurysms after introduction of the Pipeline Flex: analysis of a single-institution series of 568 cases. J Neurosurg. 2018 Dec 1;129(6):1475-1481. doi: 10.3171/2017.7.JNS171289. Epub 2018 Jan 12. PMID 29327999
- [Result] Zhang H, Zhang H, Liu J, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Luo B, Shao Q, Chang K, Zhang Q, He Y, Zhang P, Yang X, Li L, Li TX. Pipeline Embolization Device for Small and Medium Vertebral Artery Aneurysms: A Multicenter Study. Neurosurgery. 2023 May 1;92(5):971-978. doi: 10.1227/neu.0000000000002319. Epub 2022 Dec 29. PMID 36700744
- [Result] Fargen KM, Hoh BL, Welch BG, Pride GL, Lanzino G, Boulos AS, Carpenter JS, Rai A, Veznedaroglu E, Ringer A, Rodriguez-Mercado R, Kan P, Siddiqui A, Levy EI, Mocco J. Long-term results of enterprise stent-assisted coiling of cerebral aneurysms. Neurosurgery. 2012 Aug;71(2):239-44; discussion 244. doi: 10.1227/NEU.0b013e3182571953. PMID 22472556
- [Result] Wang J, Vargas J, Spiotta A, Chaudry I, Turner RD, Lena J, Turk A. Stent-assisted coiling of cerebral aneurysms: a single-center clinical and angiographic analysis. J Neurointerv Surg. 2018 Jul;10(7):687-692. doi: 10.1136/neurintsurg-2017-013272. Epub 2017 Nov 16. PMID 29146831
- [Result] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1046-e1081. doi: 10.1161/CIR.0000000000000624. Epub 2018 Nov 10. No abstract available. PMID 30565953
- [Result] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Result] Dawson LP, Lum M, Nerleker N, Nicholls SJ, Layland J. Coronary Atherosclerotic Plaque Regression: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Jan 4;79(1):66-82. doi: 10.1016/j.jacc.2021.10.035. PMID 34991791
- [Result] Diomede L, Albani D, Sottocorno M, Donati MB, Bianchi M, Fruscella P, Salmona M. In vivo anti-inflammatory effect of statins is mediated by nonsterol mevalonate products. Arterioscler Thromb Vasc Biol. 2001 Aug;21(8):1327-32. doi: 10.1161/hq0801.094222. PMID 11498461
- [Result] Wagner AH, Kohler T, Ruckschloss U, Just I, Hecker M. Improvement of nitric oxide-dependent vasodilatation by HMG-CoA reductase inhibitors through attenuation of endothelial superoxide anion formation. Arterioscler Thromb Vasc Biol. 2000 Jan;20(1):61-9. doi: 10.1161/01.atv.20.1.61. PMID 10634801
- [Result] Qiao L, Wang S, Jia Q, Bian J, Fan Y, Xu X. Clinical efficacy and safety of statin treatment after carotid artery stenting. Artif Cells Nanomed Biotechnol. 2019 Dec;47(1):3110-3115. doi: 10.1080/21691401.2019.1645149. PMID 31352800
- [Result] Tentzeris I, Rohla M, Jarai R, Farhan S, Freynhofer MK, Unger G, Nurnberg M, Geppert A, Wessely E, Wojta J, Huber K. Influence of high-dose highly efficient statins on short-term mortality in patients undergoing percutaneous coronary intervention with stenting for acute coronary syndromes. Am J Cardiol. 2014 Apr 1;113(7):1099-104. doi: 10.1016/j.amjcard.2013.12.012. Epub 2014 Jan 14. PMID 24462073
- [Result] Lilja F, Wanhainen A, Mani K. Statin therapy after elective abdominal aortic aneurysm repair improves long-term survival. Br J Surg. 2024 Jan 3;111(1):znad383. doi: 10.1093/bjs/znad383. PMID 38198155